CLINICAL TRIAL: NCT03938207
Title: The Comprehensive Analysis of Health Records, TCM Constitution, Biomarker, and Whole-genome Sequencing Among Dry Eye Syndrome, Healthy Control, Sjögren's Syndrome and Other Inflammation Disease in Taiwan
Brief Title: Dry Eye Syndrome, Healthy Control, Sjögren's Syndrome and Other Inflammation Disease in Taiwan Biobank
Status: Not yet recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-04-009ACF
Record Dates: First submitted 2019-04-22; First posted 2019-05-06 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Dry Eye Syndrome; Sjogren's Syndrome; Healthy Control; Inflammation
Keywords: Dry eye syndrome; Sjögren's syndrome; Gene modulation; Xerophthalmia; TCM pattern; Inflammation; Healthy control
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Inflammation; Xerophthalmia | interventions — Blood Specimen Collection; Urination; Nutritional Status; Medical History Taking; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The DNA of Sjögren's syndrome patients, dry eye syndrome patients, other inflammation disease, and health subjects will take to do the DNA Exome sequencing.
  The saliva of Sjögren's syndrome patients, other inflammation disease, and health subjects will take to do the oral microbiome.
  The protein of Sjögren's syndrome patients, other inflammation disease, and health subjects will take to do the proteomics.
  The RNA of Sjögren's syndrome patients, dry eye syndrome patients, other inflammation disease, and health subjects will store to do the RNA sequencing.
  The plasma of Sjögren's syndrome patients, dry eye syndrome patients, other inflammation disease, and health subjects will store to do the cytokine detection in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Dry eye syndrome: Dry eye syndrome patients were extracted from Taiwan Biobank.
  Interventions: Diagnostic Test: Whole-genome genotyping; Diagnostic Test: Whole-genome sequencing; Diagnostic Test: TCM pattern; Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Physical examination indicators, blood, urine and biochemical function test; Diagnostic Test: Demographics, personal health behavior, living environment, dietary status, family history; Diagnostic Test: HLA typing; Diagnostic Test: Full-length 16S Amplicon Sequencing; Diagnostic Test: Epigenomic; Diagnostic Test: Metabolomics; Diagnostic Test: Environmental Toxic; Diagnostic Test: Medical Image
- Health subjects: Health subjects were extracted from Taiwan Biobank.
  Interventions: Diagnostic Test: Whole-genome genotyping; Diagnostic Test: Whole-genome sequencing; Diagnostic Test: TCM pattern; Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Physical examination indicators, blood, urine and biochemical function test; Diagnostic Test: Demographics, personal health behavior, living environment, dietary status, family history; Diagnostic Test: HLA typing; Diagnostic Test: Full-length 16S Amplicon Sequencing; Diagnostic Test: Epigenomic; Diagnostic Test: Metabolomics; Diagnostic Test: Environmental Toxic; Diagnostic Test: Medical Image
- Sjögren's syndrome: Sjogren's syndrome patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
  Interventions: Diagnostic Test: Whole-genome genotyping; Diagnostic Test: Whole-genome sequencing; Diagnostic Test: TCM pattern; Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Physical examination indicators, blood, urine and biochemical function test; Diagnostic Test: Demographics, personal health behavior, living environment, dietary status, family history; Diagnostic Test: HLA typing; Diagnostic Test: Full-length 16S Amplicon Sequencing; Diagnostic Test: Epigenomic; Diagnostic Test: Metabolomics; Diagnostic Test: Environmental Toxic; Diagnostic Test: Medical Image
- other inflammation disease: Other inflammation disease were extracted from Taiwan Biobank.
  Interventions: Diagnostic Test: Whole-genome genotyping; Diagnostic Test: Whole-genome sequencing; Diagnostic Test: TCM pattern; Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Physical examination indicators, blood, urine and biochemical function test; Diagnostic Test: Demographics, personal health behavior, living environment, dietary status, family history; Diagnostic Test: HLA typing; Diagnostic Test: Full-length 16S Amplicon Sequencing; Diagnostic Test: Epigenomic; Diagnostic Test: Metabolomics; Diagnostic Test: Environmental Toxic; Diagnostic Test: Medical Image

INTERVENTIONS:
Diagnostic Test: Whole-genome genotyping — Using Whole-genome genotyping from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease.
Diagnostic Test: Whole-genome sequencing — Using whole-genome sequencing from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: TCM pattern — We want to use TCM pattern to investigate the difference among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease.
Diagnostic Test: DNA Exome sequencing — The DNA of dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease will take to do the DNA Exome sequencing.
Diagnostic Test: Physical examination indicators, blood, urine and biochemical function test — To investigate the difference of Physical examination indicators, blood, urine and biochemical function test among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease.
Diagnostic Test: Demographics, personal health behavior, living environment, dietary status, family history — To investigate the difference among the demographics, personal health behavior, living environment, dietary status, family history of among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease.
Diagnostic Test: HLA typing — Using HLA typing from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: Full-length 16S Amplicon Sequencing — Using Full-length 16S Amplicon Sequencing from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: Epigenomic — Using Epigenomic from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: Metabolomics — Using Metabolomics from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: Environmental Toxic — Using Environmental Toxic from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.
Diagnostic Test: Medical Image — Using Medical Image from Taiwan Biobank among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences.

SUMMARY:
The comprehensive analysis of health records, TCM constitution, biomarker, and whole-genome sequencing among dry eye syndrome, healthy control, Sjögren's syndrome and other inflammation disease in Taiwan: an integrated analysis between Taiwan Biobank and Sjögren's syndrome Database

DETAILED DESCRIPTION:
Method: This study wants to apply the dataset of health records, physical examination indicators, blood biomarker, urine biomarker, biochemical biomarker, gene sequence, and metabolome from Taiwan Biobank Database to explore the difference among dry eye syndrome (DES), healthy control (HC), and other inflammation disease (ID). In addition, we want to investigate the difference among the demographics, personal health behavior, living environment, dietary status, family history, Traditional Chinese medicine (TCM) body constitution, hematology test, serum biochemical test, virus test, and urine test. We also want to use the whole-genome genotyping, whole-genome sequencing, DNA methylation, HLA typing, and metabolome to investigate the difference among the genetic variant, gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences. It could find the pathogenesis-associated candidate genes and sites, and could apply to clinical diagnosis and drug development after verification and confirmation of efficacy. Integrated the Sjögren's syndrome (SJS) database, we could explore the comprehensive analysis among DES, HC, SJS, and ID. It would provide the evidence-base medicine in TCM in the future.

Expected Results:

1. To evaluate the difference among questionnaire, physical examination indicators, blood biomarker, urine biomarker and biochemical biomarker for the DES, HC, and ID.
2. To evaluate the difference among gene copy number, single nucleotide variation, chromosomal recombination, and very low-level gene expression differences for the DES, HC, and ID.
3. To evaluate the difference among gene variation and TCM body constitution for the DES, HC, and ID.
4. To evaluate the difference among gene variation for the DES, HC, SJS, and ID.
5. To establish predicting modal and biomarker among DES.

ELIGIBILITY:
Sjögren's syndrome

Inclusion Criteria:

1. aged between 20 and 75 years
2. fulfilled the 2002 American-European Consensus Criteria for SS (AECG) Exclusion Criteria: NA

Dry eye syndrome

Inclusion Criteria:

1. aged between 20 and 75 years
2. Schirmer's test less than 10 mm/5 min Exclusion Criteria: NA

Inflammation disease

Inclusion Criteria:

1. aged between 20 and 75 years
2. Disease diagnosed with Inflammation Exclusion Criteria: NA

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Subjects
  Inclusion Criteria:
  1. aged 20 and 75 years
  2. had no chronic inflammatory illness.
  Exclusion Criteria:
  1. a history of alcohol abuse, diabetes mellitus, or major life-threatening condition
  2. pregnancy or breastfeeding
  3. abnormal findings of immune, liver, kidney, or blood function evaluations
  4. total sleeping time insufficiency less than 6 hours before one day of enrollment
  5. ever took the conventional medicine or hormone within one month
  6. ever encountered the acute illness, allergy reaction, immune, or rheumatic disease within one month.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunity-related gene expression | Five year
  To evaluate the immunity-related gene expression for Dry eye syndrome, Sjögren's syndrome and healthy control.
  DNA exome combine the GATK (Genome Analysis Toolkit) is a tool for detecting the ratio of immunity-related gene expression.
TCM pattern | Five year
  To evaluate the difference of TCM pattern between Dry eye syndrome, Sjögren's syndrome and healthy control.
  TCM pattern is a tool for detecting the constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Mao Chang, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang PY, Chen CH, Chiu YF, Lin HC, Chang CM. Dietary Habits, TCM Constitutions, and Obesity: Investigating the Protective Effects of Vegetarian Dietary Patterns in Taiwan. Healthcare (Basel). 2025 Jul 8;13(14):1641. doi: 10.3390/healthcare13141641. PMID 40724666